CLINICAL TRIAL: NCT07179263
Title: Inducing Redness Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C23036014
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Redness
MeSH Terms: conditions — Erythema | interventions — glycolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facial Test Arm (Other)
  Interventions: Other: 50% glycolic acid; Other: Tape Stripping
- Facial Control Arm (No Intervention)
- Arm Test arm (Other)
  Interventions: Other: Tape Stripping
- Arm control arm (No Intervention)

INTERVENTIONS:
Other: 50% glycolic acid — Subjects use 3 drops about 0.2g of 50% Glycolic Acid product on half face under instruction, then wait for 3 minutes and wash face by tap water. Wait for 10 minutes before measuring.
  Arms: Facial Test Arm
Other: Tape Stripping — Technician use the D100 to paste on the center of the test area and make it fit the skin more completely and evenly by pump fully cover the D100 patch for 10 seconds. Stripping on each test area until the skin change into redness. The number of stripping will be recorded.
  Arms: Arm Test arm; Facial Test Arm

SUMMARY:
This clinical study employs a single-center, split-face, randomized, and on-site controlled design to compare two methods for inducing skin redness (50% Glycolic Acid application and tape stripping) on the face and forearm in a minimum of 40 healthy female subjects. The study involves instrumental measurements (erythema index and a* value), photographic analysis, and expert clinical grading at multiple time points (baseline, 10min, 30min, 1h, 2h, and 4h after induction) to evaluate and compare the efficacy and response profiles of both irritation models.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese female whose age range from 18 to 60 years old;
2. Be in general good health and good mental state;
3. Have no any broken, scars, birthmarks and other imperfections on the test area;
4. Redness/erythema ≥ grade 2 after modelling inducing (to ensure the consistency of the baseline for comparison);
5. Haven't applied Alpha hydroxyl acid in the past 3 months;
6. Not currently be participating in any other study involving the test area (Face and Forearm);
7. Not have participated in any other study involving the test area in the past one month;
8. Be willing to read, understand and able to sign the Informed Consent Form and Photo Release From;
9. Be willing to comply with all study protocol requirements.

Exclusion Criteria:

1. Intending to get pregnant, be pregnant, be lactating, be within 6 months of delivery or be unwilling to take necessary precautions to avoid a pregnancy;
2. Having used antihistamine drugs in the past 1 week or immunosuppressants in the past 1 month;
3. Take anti-allergic drug/injections in the past 1 month;
4. Presently have allergies, allergic dermatitis or skin disease;
5. Have sensitivity or even allergy to topical products, ingredients or fragranced products;
6. Have history of allergies;
7. Have history of suffering from skin diseases (such as psoriasis, eczema, psoriasis, skin cancer, etc.);
8. Have used any anti-inflammatory treatment on the test area within 2 months prior to this study starting date;
9. Has a chronic medical condition that may interfere with testing (e.g., asthma, insulin-dependent diabetes, lupus, rheumatoid arthritis or other immune/auto-immune diseases);
10. Have used any scrubs or peeling product (regardless of method) or self-tanning products or oil control products in the past 3 days;
11. Have received cosmetic medical procedures on the face (such as injectable anti-wrinkle products, cosmetic surgery, tattoo removal, home light facial procedures or home use medical devices, etc.) in the past 1 month;
12. Have excessive sun exposure or ultraviolet light in the past 1 month;
13. Have applied ortho-hydroxybenzoic acid, hydroquinone in the past 3 months; or used prescriptions (such as antibiotic, retinoids, alpha hydroxyl acid and steroid), oral contraceptives (such as Diane 35®，Jasmine®， Holgyeme®，Syndi 35®，Regulon®);
14. Avoid providing emergency contact;
15. Subjects that are not compliant to the selection criteria or not proper for participation as determined by Principal Investigator;
16. An employee of the cosmetic companies or Shanghai China-Norm Quality technical service Co., Ltd.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Change in erythema index by Mexameter® MX 18 ( | From baseline to 4-hour after inducing
Change in a* value by Chromameter CM26dG | From baseline to 4-hour after inducing
  The a*value is a parameter in the CIELAB color space (also known as Lab) that quantifies a color's position along the red-green axis .
Facial Erythema Severity via VISIA-CRP Imaging | From baseline to 4-hour after inducing
Forearm Erythema Intensity via Cross-Polarized Light Imaging | From baseline to 4-hour inducing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided